CLINICAL TRIAL: NCT06179693
Title: AIMN Multicenter Study: Staging of Lymphomas Using PET/CT
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Chiti Arturo, Professor in Diagnostic Imaging and Radiotherapy Faculty of Medicine and Surgery, Vita-Salute San Raffaele University Director, Department of Nuclear Medicine, IRCCS Ospedale San Raffaele, IRCCS San Raffaele
Other Study IDs: 34/2008/O/OSS
Record Dates: First submitted 2023-12-01; First posted 2023-12-22 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Diagnostic accuracy — As per standard procedure, patients will undergo FDG PET. Following the PET exam it will be acquired a standard CT with intravenous contrast medium, using the CT tomograph inserted inside the PET one.

SUMMARY:
In recent years, the introduction of PET/CT tomographs (which have now almost completely replaced tomographs equipped with PET alone), has allowed a significant increase in diagnostic accuracy in the majority of tumors. However, in order to reduce the radiation doses, administering CT images are acquired for patients at a low dose (generally 60mA 120kV) without the use of contrast agents. This prudential attitude, however, makes it essential to carry out "diagnostic" CT investigations which, at the end of the diagnostic process It leads to an increase in the dose administered for the patient rather than to savings.

This study aims to evaluate the possible advantages in diagnostic, economic and quality of life terms of PET/CT performed with diagnostic CT with intravenous contrast medium, with the aim of benefiting the neoplastic patient in the diagnostic process by optimizing (from a temporal and dosimetric point of view ) the diagnostic procedures to which it is subjected.

It is expected that the integrated PET/CT procedure can facilitate the process of staging the neoplasm and that this procedure can have a positive impact on the patient's quality of life while also reducing the costs incurred in terms of time and money.

ELIGIBILITY:
Inclusion Criteria:

* Established lymphoma (non-Hodgkin's lymphoma and Hodgkin's disease) being staged;
* Performing the PET/CT examination within two weeks of diagnosis and before treatment;
* Signing of the Informed Consent.

Exclusion Criteria:

* patients <18 years;
* Patients who have not signed the Informed Consent;
* Execution of previous anti-inflammatory or anti-inflammatory therapies in the 4 weeks preceding the PET exam.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with malignant lymphoma subjected to diagnostic examination by PET/CT with contrast medium in a single session, instead of on two different dates, as occurs in normal clinical practice.
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2009-10-07 (Actual); Primary Completion 2011-02-24 (Actual); Study Completion 2011-02-24 (Actual)

PRIMARY OUTCOMES:
PET/CT with contrast medium in a single session to diagnosis of patients with malignant limphoma. | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Irccs San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No